CLINICAL TRIAL: NCT02522572
Title: Quantitating the Impact of Plerixafor Alone or in Combination With Bortezomib on Plasma Cell Mobilization and the Subsequent Impact on HLA Antibody Levels
Brief Title: Quantitating the Impact of Plerixafor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E. Steve Woodle (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor-Investigator, E. Steve Woodle, Director, Solid Organ Transplantation, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Mozobil Sanofi
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Transplants and Implants
Keywords: Renal Transplantation; Desensitization; plerixafor; bortezomib
MeSH Terms: interventions — plerixafor; Bortezomib; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): 4 doses of plerixafor and plasmapheresis
  Interventions: Drug: plerixafor; Other: plasmapheresis
- Group B (Experimental): 4 doses of plerixafor, 1 dose of bortezomib, and plasmapheresis
  Interventions: Drug: plerixafor; Drug: Bortezomib; Other: plasmapheresis
- Group C (Experimental): 6 doses of plerixafor, 2 doses of bortezomib, and plasmapheresis
  Interventions: Drug: plerixafor; Drug: Bortezomib; Other: plasmapheresis

INTERVENTIONS:
Drug: plerixafor — Plerixafor will be dosed subcutaneously and administered based on group assignment.
  Other Names: Mozobil
Drug: Bortezomib — Bortezomib will be given via IV push over 3-5 seconds and administered based on group assignment.
  Other Names: Velcade
  Arms: Group B; Group C
Other: plasmapheresis — Plasmapheresis will be administered based on group assignment.

SUMMARY:
The primary objective of this study is to conduct a proof of concept pilot study that will provide a preliminary evaluation of the safety of plerixafor alone or in combination with bortezomib on plasma cell mobilization, Human Leukocyte Antigen (HLA) antibody levels and toxicity profile in sensitized patients awaiting kidney transplantation.

The secondary objective of this study is to conduct additional analyses of the study regimen on HLA antibody levels using multiple different assays and statistical analysis.

DETAILED DESCRIPTION:
The investigators have previously demonstrated that proteasome inhibition (with bortezomib) provides effective antihumoral therapy for antibody-mediated rejection (AMR) and for desensitization in kidney transplant recipients and candidates. These studies have also demonstrated that plasma cell populations exhibit significant heterogeneity. Newly produced plasma blasts and plasma cells, whether from a primary or anamnestic immunologic response, during an acute AMR, are very sensitive to proteasome inhibitor-based therapy. Of the plasma cell populations we have examined, those that demonstrate the greatest degree of resistance to proteasome inhibitor therapy are those that reside within bone marrow niches. These long lived bone marrow niche resident plasma cell (LLBMNRPC) populations demonstrate a significant degree of resistance to bortezomib therapy. This concept of plasma cell niche providing long term survival signals is supported by substantial literature from murine models. A number of signals are involved that derive from the plasma cell niche which are thought to contribute to long lived plasma cell survival including CXC-chemokine receptor 4 (CXCR4)/chemokine (C-X-C motif) ligand 12 (CXCL12) interactions, Interleukin-6 (IL-6), B cell activating factor (BAFF), and cluster of differentiation 44 (CD44). In addition, a number of cells have been demonstrated to be involved in the plasma cell niche in either human or murine models, including eosinophils, osteoclasts, bone marrow reticular cells, amongst others.

Interruption of CXCR4/CXCL12 interactions with plerixafor has been used to induce cluster of differentiation 34+ (CD34+) bone marrow stem cell mobilization into the peripheral blood. Since the CXCR4/CXCL12 interaction is also thought to be responsible for plasma cells homing to the bone marrow niche, it has been hypothesized that plerixafor may also provide systemic mobilization of bone marrow niche resident plasma cells, or alternatively, may induce a local mobilization from the bone marrow niche of plasma cells. Given that previous studies have indicated that mobilization of long lived plasma cells is thought to result in short term (less than 72 hour) survival of long lived plasma cells, this represents a significant potential for enhancement of proteasome inhibitor-based plasma cell targeting therapies. Indeed, a previous abstract from the oncology literature has provided preliminary evidence that combined plerixafor and bortezomib therapy may be of use in mobilizing the malignant myeloma cell from its bone marrow niche, thereby enhancing sensitivity to bortezomib.

The purpose of the proposed study is to conduct a proof of concept and preliminary safety evaluation of plerixafor alone and also combined therapy with plerixafor and bortezomib. The investigators have prospectively conducted a meticulous assessment of bortezomib-related toxicities in both the transplant recipient AMR and the transplant candidate desensitization populations and recently published this in Transplantation. This experience, which now includes over 100 treated patients, indicates that the toxicity profile of bortezomib is quite comparable to that which is observed in the myeloma population. The investigators' preliminary analysis of plerixafor and bortezomib based toxicities demonstrates that there is no significant degree of overlap in the toxicities and no significant reasons to have concerns regarding combinatorial toxicities a priori.

The investigators' extensive phase I/II study of bortezomib-based desensitization with and without rituximab-based memory B-cell depletion and/or plasmapheresis has provided a substantial experience as a first line approach for first generation plasma cell targeted therapies for desensitization in kidney transplant candidates. The current proposal is the first in the initiation of second generation plasma cell targeting protocols which have substantial potential for applications beyond kidney transplant candidates. These types of regimens may also lend themselves to AMR and desensitization in kidney transplant recipients and also in heart and other solid organ transplant recipients. It is also possible that such second generation plasma cell targeted protocols may also be of use for desensitization in kidney transplant, heart transplant, and other solid organ transplant populations. Finally, these plasma cell targeted therapies may also be of use in autoimmune diseases where autoantibodies are thought to represent a major pathogenetic factor.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between 18 and 65 years of age (inclusive) with end-stage renal disease awaiting kidney transplantation.
2. Patient with eligible living donor will have: donor specific antibody (DSA) against living donor of >5,000 mean fluorescence intensity (MFI) or a positive T or B cell flow cytometry crossmatch.
3. Patient that is on the kidney transplant waiting list awaiting a deceased donor transplant and has an immunodominant antibody (iAb) of >8,000MFI or has a current or peak calculated panel reactive antibody (cPRA) >20%.
4. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
5. Female subject is either postmenopausal for at least 1 year prior to initiation of study treatment, is surgically sterilized, or if of childbearing potential, agrees to practice 2 effective methods of contraception from the time of signing the informed consent form through 3 months after the last dose of plerixafor and/or bortezomib, or agrees to completely abstain from heterosexual intercourse. Women of childbearing potential must have a negative serum pregnancy test within the last 48 hours prior to receiving study medication.
6. Male subjects, even if surgically sterilized (i.e. status post-vasectomy) must agree to 1 of the following effective contraception through 3 months after end of study.
7. Review of pre-transplant medical clearance by the patient's transplant nephrologist to assure the patient is medically acceptable for study entry.
8. Cardiac evaluation by transplant nephrologist with clearance documented in writing to participate in the study.

Exclusion Criteria:

1. Known hypersensitivity to bortezomib, boron or mannitol, plerixafor or any of its components.
2. Actual body weight exceeds 175% of ideal body mass.
3. Subjects judged by the investigator to be at significant risk of failing to comply with the requirements of the protocol or unable to cooperate or communicate with the investigator.
4. Abnormal electrocardiogram (ECG) with clinically significant ventricular arrhythmias or other conduction abnormality that in the opinion of the investigator warrants exclusion of the subject from the trial.
5. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix A), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
6. Patient has Grade 2 peripheral neuropathy by Common Toxicity Criteria for Adverse Effects (CTCAE) criteria within 14 days before enrollment.
7. Patients with an absolute neutrophil count < 1,000/mm3 or platelet count < 75,000/mm3 within 30 days of consent.
8. Patient has received other investigational drugs within 14 days prior to initiation of study treatment.
9. Receipt of a live vaccine within 4 weeks prior to initiation of study treatment.
10. Received blood transfusions within 30 days prior to trial entry.
11. Serious medical (other than renal disease) or psychiatric illness likely to interfere with participation in this clinical study.
12. Patients who are anti-HIV-positive, anti-Hepatitis C Virus (HCV) positive with a detectable viral load, or HBsAg-positive on testing performed within one year of consent.
13. History of malignancy within the past 5 years that is not considered to be cured, with the exception of localized basal cell carcinoma of the skin (excised ≥ 2 years prior to randomization).
14. Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin > 1.5 times upper limit of normal (ULN)) on testing performed within 30 days of consent.
15. Patients with current or severe systemic infections.
16. Pregnant or nursing (lactating) women and women who might become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in immunodominant Donor Specific Antibody (iDSA) [highest titer DSA (MFI)] and/or immunodominant antibody (iAb) | Up to 44 days

CONTACTS AND LOCATIONS:
Overall Officials: Ervin S Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio